CLINICAL TRIAL: NCT03295552
Title: Decitabine Plus Carboplatin in the Treatment of Metastatic Triple Negative Breast Cancer
Brief Title: Decitabine Plus Carboplatin in the Treatment of Metastatic TNBC
Acronym: DETECT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow enrollment.
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Kunwei Shen, Professor, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RJBC1701
Record Dates: First submitted 2017-09-20; First posted 2017-09-28 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Breast Neoplasm
Keywords: decitabine; triple negative breast cancer; carboplatin; metastatic
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms; Neoplasm Metastasis | interventions — Decitabine; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DC (Experimental): DNA demethylating agent decitabine plus carboplatin
  Interventions: Drug: Decitabine; Drug: Carboplatin

INTERVENTIONS:
Drug: Decitabine — decitabine 7mg/m2, d1-d5, q3w
Drug: Carboplatin — carboplatin AUC = 6, d6, q3w

SUMMARY:
To evaluate the effect of novel DNA demethylating agents in the treatment of metastatic TNBC

ELIGIBILITY:
Inclusion Criteria:

* Female aged between 18 years and 70 years old.
* Pathologically confirmed metastatic triple negative breast cancer (TNBC). Paraffin-embedded tissue were available from metastatic or primary sites to confirm its TNBC status or for further translational research. TNBC was defined as ER-, PR-, and HER2-.
* Metastatic TNBC should not be treated with more than 1-line for metastatic disease.
* Patients can not be treated with carboplatin in the metastatic setting.
* For patients received carboplatin treatment in the adjuvant setting, they should have at least one year disease interval between last dosage of carboplatin and trial recruiting.
* Patients had at least one measurable lesion according to RECIST criteria version 1.1.
* ECOG Performance Status (PS) of 0-1.
* Adequate liver and renal organ function.
* Dated and signed IEC/IRB-approved informed consent.

Exclusion Criteria:

* More than 1 one therapy for metastatic TNBC, Patients may receive bisphosphonates and other therapies to treat bone metastases.
* Less than four weeks since last radiotherapy.
* Pregnancy or lactation or unwillingness to use adequate method of birth control.
* Active or uncontrolled infection.
* Hypersensitivity to carboplatin or decitabine
* Male breast cancer.
* Treated with any DNA demethylating agents
* Young patients with pregnancy or lactation or unwillingness to use adequate method of birth control.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Overall response rate | At the end of Cycle 6 (each cycle is 21 days)
  Partial response (PR) + complete response (CR) rate

CONTACTS AND LOCATIONS:
Overall Officials: Kunwei Shen, MD, Principal Investigator — Ruijin Hospital, Shanghai Jiaotong Univeristy School of Medicine; Min Lu, PHD, Principal Investigator — Ruijin Hospital, Shanghai Jiaotong Univeristy School of Medicine
Locations (1):
- Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided